CLINICAL TRIAL: NCT06259084
Title: Study to Detect the Predictive Capacity of a Composite Biological Marker in the Success of Embryonic Implantation in Fertilization Treatments in Vitro (IVF): Seedchrony Pilot.
Brief Title: Study to Estimate Seedchrony's Predictive Capacity in the Success of Embryo Implantation.
Acronym: Seedchrony02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manina Medtech (Industry)
Collaborators: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: T-015-004
Record Dates: First submitted 2024-01-21; First posted 2024-02-14 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Infertility
Keywords: embryo transfer; embryo implantation; endometrial preparation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Measurement (Experimental): Intrauterine biomarker will be measured twice in all enrolled patients during the frozen embryo transfer cycle: on the day before embryo transfer and on the day of embryo transfer.
  Interventions: Device: Seedchrony

INTERVENTIONS:
Device: Seedchrony — The seedchrony probe is coupled to the transfer catheter. When the transfer catheter is placed inside the uterus, the probe measures the biomarker concentraction in the fluid entering the catheter. The measurements last two minutes.

SUMMARY:
In Vitro Fertilization (IVF) success is below 40%, with Embryo Transfer the leading cause of IVF failure. This clinical investigation aims to evaluate if the levels of an intrauterine biomarker dissolved in the uterine fluid (alone or as a complex biological marker) can predict the outcome of embryo transfer.

DETAILED DESCRIPTION:
Seedchorny02 is an exploratory study, with blind evaluation by third parties, in a single center and without influencing clinical practice. The goal of this investigation is to evaluate if the levels of an intrauterine biomarker that is dissolved in the endometrial fluid can predict the outcome of embryo transfer, when measured the day before or on the day of embryo transfer.

80 IVF volunteers in a frozen embryo transfer cycle with high-quality day-five blastocysts are expected to be recruited. For intrauterine measurement, the investigational device Seedchrony RUO 02 will be used. Seedchorny RUO 02 has a microsensor integrated into the transfer catheter to measure the biomarker level in the uterine fluid entering the transfer catheter. Other patients' clinical variables and IVF cycle parameters (hormonal levels, ultrasound parameters, embryo quality grades, and transfer protocol) will also be collected.

Primary variable: Relationship between intrauterine dissolved biomarker concentration (alone or as a complex biological marker) and the outcome of the embryo transfer.

Notes: The intrauterine biomarker concentration is measured twice: the day before the transfer and on the transfer day. Complex biological marker refers to combining the concentration of the biomarker on both days and/or with other clinical variables of the patient/embryo.

The outcome of the embryo transfer is evaluated as:

Chemical pregnancy: positive pregnancy test (blood hGC detection); Clinical pregnancy confirmed by ultrasound at week six (detected gestational sac); Ongoing pregnancy at week eight, confirmed by ultrasound at week eight (detected gestational sac and heartbeat).

ELIGIBILITY:
Inclusion Criteria:

* First IVF cycle patients
* Patients who sign the informed consent form
* Patients between 18 and 37 years old.
* Patients BMI ≤ 30
* Patients who have frozen blastocysts of good quality (grade A or B)
* Patients with negative vaginal and endocervical cultures
* Patients with an antimullerian hormone level greater than 1 ng/mL.
* IVF patients with an endometrial thickness greater than 7mm with trilaminar pattern on the day of the pre-progesterone visit.
* And who meets one of these conditions:

  1. Not having had a previous embryo transfer.
  2. Have failed only one embryo transfer

Exclusion Criteria:

* Patients with seminal data of the couple with severe oligozoospermia (sperm concentration <1 million sperm per ml) or azoospermia (absence of sperm in the ejaculate)
* Patients diagnosed with at least one of the following uterine pathologies: endometriosis, cancer, malformations, untreated polyps, or submucous fibroids.
* Patients diagnosed with at least one of the following medical pathologies: Polycystic ovary syndrome (PCOS), insulin-dependent diabetes mellitus, Cushing's syndrome, uncorrected thyroid dysfunction, hepatic and/or renal insufficiency, a pathology that contraindicates ovarian stimulation and/or gestation, antiphospholipid syndrome, and autoimmune disease.
* Patients who are currently taking any medication other than contraceptive treatments, which may interfere with fertility or menstrual cycle regulation.
* Evidence of drug, tobacco, or alcohol abuse or dependence according to medical history or information provided by the patient.
* Inadequate understanding (oral and written) of the Spanish language.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-07-05 (Estimated)

PRIMARY OUTCOMES:
Intrauterine biomarker concentration on the day before embryo transfer | one day
  The Seedchrony probe is coupled to the transfer catheter and placed in the uterine cavity. The probe measures the biomarker concentration in the fluid entering the catheter.
Intrauterine biomarker concentration on the embryo transfer day | one day
  The Seedchrony probe is coupled to the transfer catheter and placed in the uterine cavity. The probe measures the biomarker concentration in the fluid entering the catheter.

SECONDARY OUTCOMES:
Biochemical Pregnancy | 10-14 days after embryo transfer
  Biochemical Pregnancy outcome will be measured using a serum pregnancy test at 10-14 days after embryo transfer. Results will be record as positive or negative.
Clinical Pregnancy | 4 weeks after embryo transfer
  Clinical Pregnancy outcome will be assessed by ultrasound at post-transfer week 4. Results will be record as positive or negative.
Ongoing Pregnancy | 6 weeks after embryo transfer
  Ongoing Pregnancy outcome will be assessed by ultrasound at post-transfer week 6. Results will be record as positive or negative.
User experience and device safety in the clinical environment | 12 months
  End-user experience and feedback with clinicians' satisfaction questionnaire. Report of events regarding incorrect device handling, dropping, sensor breakage, erroneous readings, and device and software failures.
Evaluate the patient's experience during measurements. | two days (day before embryo transfer and on the transfer day)
  Visual Analog Scale (VAS) will be used to measure patients' pain and discomfort during measurements. Patients will be asked to rate their experience by making a mark along a line from 1 "no pain" to 10 "worst imaginable pain or discomfort". The distance from the starting point to the mark provides a quantitative measurement of the patient's experience.

CONTACTS AND LOCATIONS:
Overall Officials: Melchor Carbonell, Dr., Principal Investigator — Hospital Universitario Vall d'Hebron Passeig de la Vall d'Hebron 119-129. 08035 Barcelona
Locations (1):
- Vall d'Hebron Hospital, Barcelona, Other (Non US), Spain

IPD SHARING:
Plan to Share IPD: No